CLINICAL TRIAL: NCT05955742
Title: Evaluation of Postoperative Pain After Using Different Single-File Glide Path Systems: a Randomized Clinical Trial
Brief Title: Postoperative Pain After Using Different Single-File Glide Path Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Kubra Yesildal Yeter, Associate Professor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EskisehirOU-endodonti
Record Dates: First submitted 2023-07-11; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Post Operative Pain
Keywords: chronic apical periodontitis; glide path preparation; Postoperative pain; ProGlider; WaveOne Gold Glider
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Group 1: control Group 2: ProGlider Group 3: WaveOne Gold Glider
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and statistician were blind to the groups but the operator who performed all treatment procedures could not be blinded to the study group owing to the study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental): Glide path preparation with hand files.
  Interventions: Device: Control
- ProGlider (Experimental): Glide path preparation using rotational NiTi file.
  Interventions: Device: ProGlider
- WaveOne Gold Glider (Experimental): Glide path was preparation using reciprocating NiTi file.
  Interventions: Device: WaveOne Gold Glider

INTERVENTIONS:
Device: Control — The operator prepared the glide path using a #15K-type stainless-steel hand file.
  Arms: Control
Device: ProGlider — The operator prepared the glide path using the ProGlider file.
  Arms: ProGlider
Device: WaveOne Gold Glider — The operator prepared the glide path using the WaveOne Gold Glider file.
  Arms: WaveOne Gold Glider

SUMMARY:
This study aimed to evaluate postoperative pain intensity after glide-path preparation with the ProGlider (PG) and WaveOne Gold Glider (WOGG) systems in asymptomatic teeth with necrotic pulp and periapical lesions.Maxillary and mandibular molars with chronic apical periodontitis of 78 patients (age, 18-65 years) were included. The patients were randomly divided into three groups: control (n = 26), PG (n = 26), and WOGG (n = 26). All systems were used according to the manufacturer's instructions, and all root canal treatments were completed by a single operator within two sessions. Postoperative pain was assessed using a numerical rating scale (NRS) at 6, 12, 18, 24, 48, and 72 h. The intake of prescribed analgesics and abscess formation were also recorded.

DETAILED DESCRIPTION:
Pain after root canal treatment is an important complication encountered in endodontic practice, with a reported prevalence of 3%-58%. Severe pain may start even 24 to 48 h after treatment. Postoperative pain has a complex etiology, including treatment factors under the control of the clinician, microbial factors related to the contents of infected root canals, patient demographic factors (patient sex and age, among others), immunological factors, local tissue changes, and psychological factors. Debris extrusion to the periapical tissues during root canal instrumentation can significantly influence the incidence and intensity of postoperative pain. The root canal instrumentation technique may play an important role in the occurrence of postoperative pain as it can induce an acute inflammatory response following periapical extrusion of necrotic tissues, infected debris, and bacteria. Previous clinical trials have evaluated the effect of reciprocation and continuous rotation kinematics on debris extrusion and postoperative pain; however, their results are conflicting.

The glide path is defined as a straight tunnel extending from the canal orifice to the physiological apical foramen. Glide-path preparation may prevent complications of root canal instrumentation; reduce risk of instrument failure, debris extrusion, and postoperative pain; and preserve root canal anatomy, thereby reducing the risk of transportation, perforation, and step and zip formation. Many NiTi glide-path file systems of different sizes and metallurgical properties have been introduced to date. Recently, a new single glide-path file system was introduced with the aim of reducing the number of files used and simplifying glide-path instrumentation.

The effect of glide-path file systems on postoperative pain has been studied previously. However, to the best of investigators' knowledge, there are no data comparing PG and WOGG glide-path files in terms of postoperative pain in asymptomatic teeth with necrotic pulp and periapical lesions. Therefore, the purpose of this in vivo study was to evaluate the incidence and intensity of postoperative pain in asymptomatic maxillary and mandibular molars with necrotic pulp and periapical lesions after glide-path preparation with a stainless-steel K-file and PG and WOGG glide-path file systems. The null hypothesis was that there is no difference in the incidence and intensity of postoperative pain between glide-path preparation techniques.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic maxillary and mandibular first and second molars diagnosed with chronic apical periodontitis in healthy patients
* Patients between 18-65 years old
* Patients who had not taken antidepressants, sedative drugs, analgesics and/or anti-inflammatory drugs
* Patients who could understand the use of numeric rating scale (NRS) for pain.

Exclusion Criteria:

* Patients who were allergic to anesthetics and non-steroidal drugs
* Patients who use immunosuppressants
* Patients who are pregnant or breastfeeding
* Patients with systemic infections.
* Teeth with advanced periodontal disease
* Teeth with acute pain
* Teeth with calcified or resorbed canals
* Teeth with complex root canal anatomy
* Teeth with vital pulp
* Unrestorable teeth
* Presence of cracks and/or fractures
* Teeth associated with acute and chronic apical abscesses

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity following the use of different glide path preparations | 6th hour
  Postoperative pain was assessed using a numerical rating scale (NRS), The severity of pain varies between 0 to 10, in which 0 means no pain, while 10 means unbearable pain.
Postoperative pain intensity following the use of different glide path preparations | 12th hour
  Postoperative pain was assessed using a numerical rating scale (NRS), The severity of pain varies between 0 to 10, in which 0 means no pain, while 10 means unbearable pain.
Postoperative pain intensity following the use of different glide path preparations | 18th hour
  Postoperative pain was assessed using a numerical rating scale (NRS), The severity of pain varies between 0 to 10, in which 0 means no pain, while 10 means unbearable pain.
Postoperative pain intensity following the use of different glide path preparations | 24th hour
  Postoperative pain was assessed using a numerical rating scale (NRS), The severity of pain varies between 0 to 10, in which 0 means no pain, while 10 means unbearable pain.
Postoperative pain intensity following the use of different glide path preparations | 48th hour
  Postoperative pain was assessed using a numerical rating scale (NRS), The severity of pain varies between 0 to 10, in which 0 means no pain, while 10 means unbearable pain.
Postoperative pain intensity following the use of different glide path preparations | 72nd hour
  Postoperative pain was assessed using a numerical rating scale (NRS), The severity of pain varies between 0 to 10, in which 0 means no pain, while 10 means unbearable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Kubra Yesildal Yeter, Assoc. Prof., Principal Investigator — Eskisehir Osmangazi University
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Danaci Z, Yeter KY. Evaluation of Pain Following the Use of Different Single-file Glide Path Systems: A Randomized Clinical Trial. J Endod. 2024 Feb;50(2):120-128. doi: 10.1016/j.joen.2023.10.017. Epub 2023 Nov 3. PMID 37924939